CLINICAL TRIAL: NCT00501150
Title: A Prospective Implementation of an IV-oral Switch Policy to Treat Proven or Suspected Infections Due to Resistant Gram Positive Bacteria in a London Hospital Trust
Brief Title: Oral Antibiotic Treatment at Home Instead of Intravenous Treatment in Hospital for Resistant Gram Positive Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Hammersmith Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BAMK1021; 05/q0406/106
Record Dates: First submitted 2007-07-12; First posted 2007-07-13 (Estimated); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Gram-positive Bacterial Infections; Staphylococcal Infections
Keywords: linezolid; vancomycin; glycopeptides; methicillin resistant staphylococcus aureus; resistant gram positive infections
MeSH Terms: conditions — Gram-Positive Bacterial Infections; Staphylococcal Infections | interventions — Linezolid

ARMS (1):
- Patients who fulfilled the study criteria (Experimental): IV to oral switch inclusion criteria used
  1. Clinical status
     * Temperature less than 38°C for 24 hours
     * White cell count normalising
     * No unexplained tachycardia (Heart rate less than 100 beats per minute)
     * Sensitivity received (if microbiology positive)
  2. Oral absorption
     * Patient tolerates oral fluids
     * No medical problems leading to reduced oral absorption (e.g. vomiting, diarrhoea, and gastrointestinal surgery)
     * No surgical operation scheduled within next 36 hours
  IV to oral switch exclusion criteria used
  1. Continuing sepsis
     * Temperature less than 36°C or more than 38°C
     * White cell count less than 4 × 109/L or more than 12 × 109/L
     * Unexplained tachycardia (Heart rate greater than 100 beats per minute in last 12 hours)
  2. Oral route compromised
     * Vomiting or severe diarrhoea
     * Other ongoing or potential absorption problem
  Interventions: Drug: linezolid

INTERVENTIONS:
Drug: linezolid — Linezolid is an antimicrobial with activity against MRSA that can be given orally.

SUMMARY:
The main purpose of this study is to find out whether changing the hospital policy to allow switch from glycopeptide antibiotics (given by intravenous drip), to an equally effective oral antibiotic (linezolid) will enable patients who are otherwise well enough to be discharged from hospital sooner.

The secondary objectives are

1. To identify those patients who could potentially be discharged on an oral agent from those being treated with a glycopeptide, thus helping target this approach most effectively
2. To evaluate the cost involved and compare this with the costs that would have taken place if use of an oral agent and discharge had not occurred.

DETAILED DESCRIPTION:
The treatment of resistant gram positive infections remains problematic, with glycopeptides remaining the mainstay of current management. Unfortunately these can only be administered by the IV route, with no useful activity when given orally for these infections. Thus while oral flucloxacillin or ampicillin are used as follow up to IV treatment in the management of infections caused by antibiotic sensitive Staphylococcus aureus or enterococcal respectively, in the case of antibiotic resistant infections the whole course of antibiotics is usually given by the IV route. To some extent this is because there is insufficient evidence to support routine use of other oral agents and means that patients with antibiotic resistant infections stay in hospital longer than those with antibiotic sensitive infections.

Linezolid is a relatively newly available antibiotic that has been shown to be as, and in some settings more effective than glycopeptides in the treatment of resistant gram positive infections including MRSA. Unfortunately Linezolid is significantly more expensive than other currently available agents making it important to evaluate the cost benefit aspects of its use in comparison to similarly effective agents.

Switching from IV to a suitable oral alternative in the management of resistant gram positive infection could potentially result in significant saving in the duration of IV therapy and would allow patients to be discharged earlier. This would provide a significant cost benefit which in the face of Linezolids equal if not superior efficacy would justify more widespread use in order to allow suitable patients to be treated at home.

The rationale behind this study is to determine the level at which this can be implemented in an NHS teaching hospital Trust. To do this we will identify patients who could potentially benefit from early discharge on oral therapy, implement this where possible and compare the actual effect on LOS with the potential identified in the earlier cohort of patients.

We propose to prospectively assess the economic and clinical impact of switching from IV glycopeptides to oral Linezolid and implementing home treatment on oral therapy policy over an 18 month period in HHT hospitals Two senior infection specialists(a Medical Microbiologist, K Bamford and an Infectious Disease physician, A Holmes) will independently review each patient together with the study pharmacist and decide if the individual is suitable for switch to an oral agent and/or discharge using standardised criteria for decision making. Patients will be studied to assess the number of attributable bed days, line use days, ward pharmacist interventions (to trigger monitoring and adjust dose) and investigations and medical complications that accrue due to IV administration following glycopeptide prescription. The various costs to the Trust which are saved when the IV glycopeptide is switched to a suitable oral alternative and early discharge implemented will be calculated

ELIGIBILITY:
Inclusion Criteria:

1. Prescribed five or more days glycopeptide
2. Fulfil IV-oral switch criteria (see below) with likelihood of discharge within next 48 hours.

Exclusion Criteria:

1. Renal dialysis out patients
2. Suspected or proven left sided endocarditis/osteomyelitis/prosthetic infection where the prosthesis cannot be removed
3. Per-protocol prescribing in haematology (i.e. where teicoplanin is prescribed in response to failure of fever resolution in neutropenic patients without microbiological or clinical evidence of gram positive infection).
4. Age < 16 years
5. Pregnant or lactating female.
6. Other contraindication to linezolid
7. Clinically unlikely to be discharged within study period or at end of antibiotic therapy.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2005-09 (Actual); Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
To identify the percentage of patients currently prescribed IV glycopeptides who could be discharged earlier if an oral agent was used | Period between IV oral switch and discharge, at least 24 hours

SECONDARY OUTCOMES:
To estimate the number of inpatient days that could be saved | Period between IV oral switch and discharge, at least 24 hours
To identify the groups of patients most likely to be suitable for earlier discharge if an oral agent was used | Period between IV oral switch and discharge, at least 24 hours
To identify the additional number of days of IV antibiotic treatment that could be prevented by using an oral agent in hospitalised patients | Period between IV oral switch and discharge, at least 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen B Bamford, MB BCh BAO, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London, London, United Kingdom

REFERENCES:
- [Result] Desai M, Franklin BD, Holmes AH, Trust S, Richards M, Jacklin A, Bamford KB. A new approach to treatment of resistant gram-positive infections: potential impact of targeted IV to oral switch on length of stay. BMC Infect Dis. 2006 Jun 8;6:94. doi: 10.1186/1471-2334-6-94. PMID 16762061